CLINICAL TRIAL: NCT04698148
Title: Costituzione Della Biobanca Del Microbiota Intestinale e Salivare Umano: Dalla Disbiosi Alla Simbiosi
Brief Title: Establishment of the Human Intestinal and Salivary Microbiota Biobank - Gastrointestinal Diseases
Acronym: BIOMIS-Gastr
Status: Completed | Type: Observational
Sponsor: Azienda Ospedaliero-Universitaria Consorziale Policlinico di Bari (Other)
Collaborators: Istituti Tumori Giovanni Paolo II (Network); University of Bari Aldo Moro (Other); University of Salento (Other); University Of Perugia (Other); Institute of Biomembranes, Bioenergetics and Molecular Biotechnologies (Other); Catholic University of the Sacred Heart (Other)
Responsible Party: Sponsor
Other Study IDs: BIOMIS-Gastr
Record Dates: First submitted 2020-12-17; First posted 2021-01-06 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2022-01

CONDITIONS: Clostridium Difficile Infection; Multi Drug Resistant Organisms; Chronic Inflammatory Bowel Disease; Irritable Bowel Syndrome; Hepatic Encephalopathy
Keywords: Microbioma biobank; Biological human samples; Gastrointestinal disease; Meta-omics approaches; Microbiota-pathology relationship
MeSH Terms: conditions — Clostridium Infections; Irritable Bowel Syndrome; Hepatic Encephalopathy; Gastrointestinal Diseases | interventions — Surveys and Questionnaires; Independent Medical Evaluation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — faeces, saliva, blood, serum, urine, PBMC
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- CDI patients: Patients with Clostridium Difficile Infection
  Interventions: Other: Biological sample collection; Other: Questionnaire; Other: Medical examination
- MDRO patients: Patients with Multi Drug Resistant Organisms infection
  Interventions: Other: Biological sample collection; Other: Questionnaire; Other: Medical examination
- IBD patients: Patients with Chronic Inflammatory Bowel Disease
  Interventions: Other: Biological sample collection; Other: Questionnaire; Other: Medical examination
- IBS patients: Patients with Irritable Bowel Syndrome
  Interventions: Other: Biological sample collection; Other: Questionnaire; Other: Medical examination
- Hepatic Encephalopathy patients: Patients with Hepatic Encephalopathy
  Interventions: Other: Biological sample collection; Other: Questionnaire; Other: Medical examination
- healthy volunteers: healthy volunteers
  Interventions: Other: Biological sample collection; Other: Questionnaire; Other: Medical examination

INTERVENTIONS:
Other: Biological sample collection — Collection of faeces, coproculture examination, urine, saliva, PBMC and blood for biobanking, to evaluate the proteomic, metascriptomic, metabolomic, metagenomic, and metagenetic profile, and to perform routine screening. Analysis for the identification, quantification and characterization of health-promoting bacteria
Other: Questionnaire — Anamnestic questionnaire, 3-day food questionnaire, Food Frequency Questionnaire
Other: Medical examination — Blood pressure measurement, abdominal and thoracic physical examination

SUMMARY:
This is a prospective, clinical, multicentre study aimed to collect biological samples and study microbiota from subjects with Clostridium Difficile (CDI), subjects affected by Multi Drug Resistant Organisms (MDRO) infection, subjects with Chronic Inflammatory Bowel Disease (IBD), subjects with Irritable Bowel Syndrome (IBS), subjects with Hepatic Encephalopathy and from healthy volunteers. Microbiota is a complex consortium of microorganisms, located at the mucosal level (in particular intestinal, oral and vaginal) having a key role in human health and in the onset of several diseases. Microbiota alterations have been found in several diseases (gastrointestinal, metabolic, renal, oncological, gynaecological)

The study will allow to:

* Provide biological samples (faeces, saliva, blood, urine) from healthy volunteers and patients to the first Italian microbiota biobank;
* Study microorganisms using different in vitro and in vivo techniques;
* Study the link between the microbiota and the disease. This study is part of the BIOMIS project (Project Code: ARS01_01220), presented as part of the "Avviso per la presentazione di progetti di ricerca industriale e sviluppo sperimentale nelle 12 aree di specializzazione individuate dal PNR 2015-2020" and admitted to funding under the National Operational Program "Ricerca e Innovazione" 2014-2020 by directorial decree of MIUR - Department for Higher Education and Research - n. 2298 of 12 September 2018. BIOMIS includes several clinical studies that enrol patients with different pathologies to collect and store biological samples and study microbiota.

DETAILED DESCRIPTION:
The primary aim of this multicentric study is to populate the first national microbioma biobank with biological samples (fecal, salivary, urinary and blood samples) subjects suffering from selected disease (CDI, MDRO, IBD, IBS and Hepatic Encephalopathy), and healthy volunteers.

The secondary aim is the characterization of microorganisms of the biobank and study of the microbiota-pathology relationship using meta-omics, in vitro and in vivo approaches.

The study plans to enrol 225 subjects at Policlinico of Bari, University of Perugia and Policlinico Agostino Gemelli Rome, according to the inclusion/exclusion criteria. The study participation is voluntary, and the subjects have the right to withdraw from the study at any time and for any reason.

During the study, 3 visits are planned:

* Visit 0 (V0), including description of the objectives and procedures study, signature written informed consent, inclusion/exclusion criteria evaluation, medical examination (blood pressure measurement, abdominal and thoracic physical examination), filling in of the anamnestic questionnaire, delivery of the coproculture kit, delivery of kits for the collection of fecal, salivary and urinary material to be reported at Visit 1 and delivery of a 3-day food diary, to be completed autonomously in the days preceding the Visit 1.
* Visit 1 (V1) - at least 4 days after V0, including delivery of the of the collected biological material (feces, saliva, urine), and of a 3-day food diary, filling in of the new signs and symptoms anamnestic questionnaire and blood sampling by medical staff. For MDRO patients rectal swab collection.
* Telephone evaluation: administration of a "Food Frequency Questionnaire" to assess the subjects' alimentary habits.

Standard Operative Procedures (SOP) for samples storing, transport and processing will be adopted to ensure samples stability and grant results validity and quality.

Following collections, samples will be processed in different aliquots that will be used for:

* routine screening;
* storage in the first Italian human microbiote biobank (I.R.C.C.S. - Istituto Tumori "Giovanni Paolo II", Bari);
* evaluation of the proteomic, metascriptomic, metabolomic, metagenomic, and metagenetic profile;
* Evaluation of the transcriptomic profile of PBMCs of healthy subjects and subjects affected by selected pathologies and evaluation of the serum proteomic profile Furthermore, molecular characterization of pathogenic microorganisms and pathogenic biotypes (pathovars) of commensal species of subjects with selected pathologies will be conducted.

Part of the biological material will be used for animal studies on the physiopathological role of the human intestinal microbiota transplanted into mouse models of pathology and Germ-free mouse models (specific animal study protocol developed).

Also, in vitro studies on mucosal models to evaluate the interaction between the microbiota and the intestinal mucosa will be conducted.

The study foresees no more than minimal risk associated with blood sampling procedures. All the necessary measures to avoid any risks / inconveniences resulting from participation of the subject under study will be taken.

The study is compliant with Good Clinical Practice. Study protocol and all related documents have been approved by approved by the Independent Ethics Committees (IEC) of the involved clinical sites.

To ensure the protection and confidentiality of the participants' data, all study activities will be carried out in accordance with the European General Data Protection Regulation, Regulation (EU) 2016/679, which repeals Directive 95/46/EC.

ELIGIBILITY:
Inclusion Criteria:

HEALTHY VOLUNTEERS

* healthy subjects aged between 18 and 60 years
* BMI between 18.5-30
* omnivorous diet
* signature of the informed consent

PATIENTS WITH CDI

* subjects with CDI > 18 years
* Symptomatic recurrent CDI infection, diagnosed by toxin search (ELISA)
* Subjects eligible for antibiotic treatment in accordance with European guidelines
* Possibility of being subjected to the diagnostic and therapeutic procedures of the study
* Negative parasitological examination of stools for Giardia lamblia, Entamoeba histolytica / dispar, Cryptosporidium parvum, and other parasites.
* Negativity of co-culture for Salmonella spp., Shigella spp., Yersinia enterocolitica, Campylobacter, Streptococcus agalactiae, Staphylococcus aureus, enteropathogenic Escherichia coli and other microorganisms with the exception of Clostridium difficile
* Negativity of the following serological tests: HAV-IgM, HBsAg, Anti-HCV, Anti-HIV1-2, VDRL
* Signature of the informed consent

PATIENTS WITH MDRO

* Subjects > 18 years old
* Subjects colonised for MDRO diagnosed with rectal swab
* Negative parasitological faeces culture for Giardia lamblia, Entamoeba histolytica / dispar, Cryptosporidium parvum and other parasites.
* Negative faeces culture for C. difficile, Salmonella spp., Shigella spp., Yersinia enterocolitica, Campylobacter, Streptococcus agalactiae, Staphylococcus aureus, enteropathogens Escherichia coli
* Signature of informed consent.

PATIENTS WITH IBD

* Age> 18 years.
* Individuals available for scheduled visits, treatment plan, laboratory tests, lifestyle guidelines, and other study procedures.
* Subjects with a documented diagnosis of ulcerative colitis or Crohn's at least 6 months before screening.
* Signature of informed consent.

PATIENTS WITH IBS

* Subjects diagnosed with IBS according to Rome IV criteria
* Age between 18 and 60 years
* BMI between 18.5-30
* Omnivorous diet
* Signature of informed consent

PATIENTS WITH HEPATIC ENCEPHALOPATHY

* Subjects with hepatic encephalopathy
* Age between 18 and 60 years
* BMI between 18.5-30
* Omnivorous diet
* Signature of informed consent

Exclusion criteria:

Healthy volunteers

* Current or previous infectious diseases (HAV, HBV, HCV, HIV, Cytomegalovirus, Epstein-Barr virus)
* Chronic liver disease
* History of Clostridium difficile infections
* Recent (<3 months) therapy with antibiotics, immunosuppressive drugs, chemotherapy
* Chronic therapy with proton pump inhibitors
* Recent (<3 months) use of probiotics, laxatives or other aids (drugs / supplements) for the regulation of gastrointestinal activity
* Previous history of organ / tissue transplantation
* Recent onset of diarrhea
* Chronic diarrhea
* Chronic constipation
* Previous gastrointestinal surgery (eg gastric bypass)
* Recurring urinary tract infections (3 cases per year)
* Previous major acute cardiovascular diseases (myocardial infarction, stroke)
* Type 2 diabetes mellitus
* Hypertension
* eGFR (estimated glomerular filtration rate) lower than 60ml / minute and / or diagnosis of nephropathy
* Chronic gastrointestinal disorders
* Systemic inflammatory diseases
* Suspicion, clinical diagnosis or previous history of cancer (<5 years)
* Autoimmune disorders or history of chronic and systemic autoimmune disorders
* Neurodegenerative disorders
* Pregnancy and breastfeeding
* Healthcare workers
* Operators work with animals
* Psychiatric conditions that reduce protocol compliance.

Patients with CDI

* Age <18 years
* Negative detection of Clostridium difficile toxin in faeces by ELISA method
* Severe clinical condition (sepsis, severe dehydration, important co-morbidities)
* Previous i.c. total or partial colectomy
* High risk of post-colonoscopy complications
* Other causes of symptoms similar to those caused by CDI, such as other infections, inflammatory bowel diseases or irritable bowel syndrome
* Positive parasitological examination of stool for Giardia lamblia, Entamoeba histolytica / dispar, Cryptosporidium parvum, and other parasites
* Copro-culture positive for Salmonella spp., Shigella spp., Yersinia enterocolitica, Campylobacter, Streptococcus agalactiae, Staphylococcus aureus, enteropathogenic Escherichia coli and other microorganisms except for Clostridium difficile
* Positivity of the following serological tests: HAV-IgM, HBsAg, Anti-HCV, Anti-HIV1-2, VDRL
* Pregnancy or breastfeeding
* Psychiatric conditions that reduce protocol compliance

Patients with MDRO

* Subjects <18
* Subjects unable to perform or intolerant to lower endoscopy
* Subjects negative for rectal swab MDRO
* Positivity for parasitological faeces culture for Giardia lamblia, Entamoeba histolytica / dispar, Cryptosporidium parvum and other parasites.
* Positive faeces culture for C. difficile, Salmonella spp., Shigella spp., Yersinia enterocolitica, Campylobacter, Streptococcus agalactiae, Staphylococcus aureus, enteropathogens Escherichia coli.
* Subjects being treated with cyclosporine, mycophenolate or tacrolimus
* Women who are pregnant or breastfeeding
* Psychiatric conditions that reduce protocol compliance

Patients with IBD

* Subjects <18 years.
* Subjects diagnosed with not determined colitis
* Patients with significant comorbidities (sepsis, severe trauma within the last 4 weeks, NYHA class IV heart failure)
* Patients with symptoms compatible with those caused by IBD, such as infectious colitis, irritable bowel syndrome, ischemic colitis, actinic colitis.
* Subjects receiving or expected to receive cyclosporine, mycophenolate or tacrolimus within 4 weeks of the first day study visit.
* Positivity for parasitological faeces culture for Giardia lamblia, Entamoeba histolytica / dispar, Cryptosporidium parvum and other parasites.
* Positive faeces culture for C. difficile, Salmonella spp., Shigella spp., Yersinia enterocolitica, Campylobacter, Streptococcus agalactiae, Staphylococcus aureus, enteropathogens Escherichia coli.
* Patients diagnosed with primary sclerosing cholangitis.
* Women who are pregnant or breastfeeding.
* Psychiatric conditions that reduce protocol compliance

Patients with IBS

* Current or previous infectious diseases (HAV, HBV, HCV, HIV, Cytomegalovirus, Epstein-Barr virus)
* Chronic liver disease
* History of C. difficile infections
* Recent (<3 months) therapy with antibiotics, immunosuppressive drugs, chemotherapy
* Chronic therapy with proton pump inhibitors
* Previous history of organ / tissue transplantation
* Previous gastrointestinal surgery (eg gastric bypass)
* Recurrent urinary tract infections (3 cases per year)
* Previous major acute cardiovascular diseases (myocardial infarction, stroke)
* Type 2 diabetes mellitus
* eGFR lower than 60ml / minute and / or diagnosis of nephropathy
* Systemic inflammatory diseases
* Suspicion, clinical diagnosis or previous history of cancer (<5 years)
* Autoimmune disorders or history of chronic and systemic autoimmune disorders
* Neurodegenerative disorders
* Pregnancy and breastfeeding
* Psychiatric conditions that reduce protocol compliance.

Patients with hepatic encefalopathy

* History of C. difficile infections
* Chronic therapy with proton pump inhibitors
* Previous history of organ / tissue transplantation
* Recent emergence of diarrhea
* Chronic diarrhea
* Previous gastrointestinal surgery (eg gastric bypass)
* Recurring urinary tract infections (3 cases per year)
* Previous major acute cardiovascular diseases (myocardial infarction, stroke)
* Type 2 diabetes mellitus
* eGFR lower than 60ml / minute and / or diagnosis of nephropathy
* Systemic inflammatory diseases
* Suspicion, clinical diagnosis or previous history of cancer (<5 years)
* Autoimmune disorders or history of chronic and systemic autoimmune disorders
* Pregnancy and breastfeeding
* Psychiatric conditions that reduce protocol compliance

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Subjects with C. Difficile (CDI), subjects affected by Multi Drug Resistant Organisms (MDRO) infection, subjects with Chronic Inflammatory Bowel Disease (IBD), subjects suffering from Irritable Bowel Syndrome (IBS) and subjects with Hepatic Encephalopathy attending one of the clinical centres involved in the study.
  Healthy volunteers will be recruited by invitation. Enrolled subjects must not have any family relationship and hierarchical subordination with the hospitals in which biological samples will be collected.
Sampling Method: Non-Probability Sample
Enrollment: 225 (Actual)
Dates: Start 2021-02-08 (Actual); Primary Completion 2022-05-10 (Actual); Study Completion 2022-05-10 (Actual)

PRIMARY OUTCOMES:
Biological samples collection for establishment of the first National Microbiome Biobank | through study completion, an average of 1 year
  Recruitment of 225 subjects (CDI, MDRO, IBD, IBS, Hepatic Encephalopathy patients and healthy volunteers) to collect biological samples for establishment of the first National Microbiome Biobank

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Losurdo, MD, Principal Investigator — Azienda Ospedaliera Universitaria Consorziale Policlinico di Bari
Locations (3):
- Italy (3):
  - Azienda Ospedaliera Universitaria Policlinico di Bari - Sezione di Malattie dell'Apparato Digerente, Endoscopia e Trapianto di Fegato (D.E.T.O.), Bari
  - Università degli Studi di Perugia - Dipartimento di Medicina, Perugia
  - Centro Malattie Apparato Digerente - CEMAD, Policlinico Universitario Agostino Gemelli IRCCS - Università Cattolica del Sacro Cuore, Roma

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aira A, Feher C, Rubio E, Soriano A. The Intestinal Microbiota as a Reservoir and a Therapeutic Target to Fight Multi-Drug-Resistant Bacteria: A Narrative Review of the Literature. Infect Dis Ther. 2019 Dec;8(4):469-482. doi: 10.1007/s40121-019-00272-7. Epub 2019 Oct 25. PMID 31654298
- [Background] Rivera-Flores R, Moran-Villota S, Cervantes-Barragan L, Lopez-Macias C, Uribe M. Manipulation of microbiota with probiotics as an alternative for treatment of hepatic encephalopathy. Nutrition. 2020 May;73:110693. doi: 10.1016/j.nut.2019.110693. Epub 2019 Dec 6. PMID 32065881
- [Background] Yoon YK, Suh JW, Kang EJ, Kim JY. Efficacy and safety of fecal microbiota transplantation for decolonization of intestinal multidrug-resistant microorganism carriage: beyond Clostridioides difficile infection. Ann Med. 2019 Nov-Dec;51(7-8):379-389. doi: 10.1080/07853890.2019.1662477. Epub 2019 Sep 13. PMID 31468999
- [Background] Ni J, Wu GD, Albenberg L, Tomov VT. Gut microbiota and IBD: causation or correlation? Nat Rev Gastroenterol Hepatol. 2017 Oct;14(10):573-584. doi: 10.1038/nrgastro.2017.88. Epub 2017 Jul 19. PMID 28743984
- [Background] Rajilic-Stojanovic M, Jonkers DM, Salonen A, Hanevik K, Raes J, Jalanka J, de Vos WM, Manichanh C, Golic N, Enck P, Philippou E, Iraqi FA, Clarke G, Spiller RC, Penders J. Intestinal microbiota and diet in IBS: causes, consequences, or epiphenomena? Am J Gastroenterol. 2015 Feb;110(2):278-87. doi: 10.1038/ajg.2014.427. Epub 2015 Jan 27. PMID 25623659